CLINICAL TRIAL: NCT01617265
Title: Prevention of Oversedation in Intensive Care Patients Under Mechanical Ventilation : the AWARE Multicentric Randomized Trial
Brief Title: Study of a Strategy to Prevent Oversedation in Intensive Care Patients Under Mechanical Ventilation
Acronym: AWARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Society for Intensive Care (Other)
Collaborators: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SRLF-TG-1-AWARE; 2011-004246-18 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: ICU Patients Requiring Invasive Mechanical Ventilation
Keywords: intensive care; mechanical ventilation; sedatives; morphinics; oversedation; mortality; midazolam; propofol; pain; agitation
MeSH Terms: conditions — Pain; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prevention of oversedation group (Experimental): In this arm sedation and analgesia will be administered according to a bundle of measures aimed at limiting oversedation, including repeated assessment of patients needs and graduate therapeutic response to control pain, discomfort, poor synchrony with the ventilator and agitation. The therapeutic options include non hypnotic anxiolytics, repeated intravenous (IV) hypnotics boluses, short-duration (6 hours) IV hypnotics infusion and round the clock IV hypnotics infusion.
  Interventions: Procedure: Clinical Procedure to Prevent Oversedation
- Conventional sedation group (Active Comparator): In this arm, sedation will be administered according to the usual practices in each participating center.
  Interventions: Procedure: Usual sedation practice

INTERVENTIONS:
Procedure: Clinical Procedure to Prevent Oversedation — Sedation and analgesia will be administered according to a bundle of measures aimed at limiting oversedation, including repeated assessment of patients needs and graduate therapeutic response to control pain, discomfort, poor synchrony with the ventilator and agitation. The therapeutic options include non hypnotic anxiolytics, repeated IV hypnotics boluses, short-duration (6 hours) IV hypnotics infusion and round the clock IV hypnotics infusion.
  Arms: Prevention of oversedation group
Procedure: Usual sedation practice — Sedation and analgesia will be administered according to the usual practices in each participating center.
  Arms: Conventional sedation group

SUMMARY:
The purpose of the present study is to determine whether administration of sedation according to a strategy including a bundle of measures to prevent oversedation is associated with a reduction in mortality of intensive care unit patients requiring mechanical ventilation, compared to administration of sedation according to usual practices.

DETAILED DESCRIPTION:
In intensive care unit (ICU) patients receiving mechanical ventilation (MV), potent hypnotics and morphinics are frequently administered to increase synchrony with the ventilator, control agitation and decrease discomfort and pain due to the tracheal tube, bed ridding, painful condition and diagnostic or therapeutic procedures.

However, administration sedatives or morphinics is often excessive and may result in deep and prolonged alteration of consciousness, delayed weaning from MV and prolonged MV. and exposes the patient to a higher risk of ventilator-associated pneumonia, ICU delirium and neuromuscular weakness at awakening.

The present randomized multicenter study will compare the day-90 mortality of a group of patients receiving conventional sedation to the mortality of a group of patients receiving sedation administered according to an algorithm aimed to prevent oversedation to the mortality. The algorithm is built on a graduate therapeutic response to increasingly intense symptoms of discomfort, pain, ventilator dyssynchrony and agitation, and includes the use of analgesics, non hypnotic benzodiazepines, neuroleptics, repeated intravenous (IV) boluses of hypnotics and short duration (6 hours) IV hypnotic infusions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Admission to ICU with expected mechanical ventilation duration > 48 hrs
* Mechanical ventilation in ICU for less than 12 hours
* Information provided to the patient or proxy

Exclusion Criteria:

* ICU Admission after cardiac arrest
* Acute or chronic neuromuscular disease
* Tracheotomy on ICU admission
* Acute cerebral injury with intracranial hypertension requiring continuous IV sedation with or without neuromuscular blockade
* Status epilepticus
* Treatment withdrawal decision
* Pregnancy, breast feeding
* Concurrent participation in another interventional study requiring a change in usual practice of sedation or mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Day-90 mortality | Mortality at Day 90 after randomization

SECONDARY OUTCOMES:
Mortality at Day 28 | at day 28
Hospital mortality | at hospital discharge, up to day 90
1-yr mortality | at 1 yr
Mechanical ventilation duration | From onset of mechanical ventilation to day 28
Days alive with no mechanical ventilation | From ICU admission up to day 28
Occurence of ventilator-associated pneumonia | During mechanical ventilation duration, up to day 28
Use of non-invasive ventilation after extubation | From extubation to ICU discharge up to day 28
Duration of ICU stay | From ICU admission to ICU discharge or death in ICU, up to day 90
ICU confusion | From Day 1 to 7, and at day 14, 21 and 28
  Number of patients alive, awaken, and free of ICU-delirium assessed on the CAM-ICU
Proximal muscle weakness | from day 1 to 7, and at day 14, 21 and 28
  Number of patients alive, awaken, cooperative and free of proximal muscle weakness
Functional, cognitive and psychological status | At day 90 and 1 year
  Functional status (measured on the Barthel scale), depression (measured on the Hospital Anxiety & Depression Scale), Posttraumatic stress disorder (measured on the Impact of Event Scale), Quality of Life (measured on the SF-36) and patient living location
Time to weaning onset | Time from mechancial ventilation initiation to first spontaneous breathing trial, up to day 28
Number of patients requiring tracheotomy | During ICU stay, up to day 28
First sitting in chair | During ICU stay, up to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DE JONGHE, MD, Study Chair — French Society of Intensive Care
Locations (43):
- France (43):
  - Hôpital Saint-Esprit, Agen
  - CHU d'Angers, Angers
  - Hopital Privé d'Antony, Antony
  - CH d'Argenteuil, Argenteuil
  - CH Germon et Gauthier, Beuvry
  - Hopital Avicenne, Bobigny
  - Hopital St-Andre, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - CHRU de la Cavale Blanche, Brest
  - Hopital Antoine Beclere, Clamart
  - CH Sud Francilien, Corbeil-Essones
  - CHU Henri Mondor, Créteil
  - Hopital Raymond Poincare, Garches
  - CHD Les Oudairies, La Roche-sur-Yon
  - CH de Versailles, Le Chesnay
  - CHU Kremlin-Bicetre, Le Kremelin-Bicetre
  - Hopital Roger Salengro, Lille
  - CH St-Joseph St-Luc, Lyon
  - Groupe Hospitalier Edouard Herriot, Lyon
  - CHU Marseille Hopital Nord, Marseille
  - Hopital de la Timone, Marseille
  - CH de Meaux, Meaux
  - Hopital Notre-Dame de Bon Secours, Metz
  - CH Princesse Grace, Monaco
  - GHIRM, Montfermeil
  - Hopital Laennec, Nantes
  - Hopital l'Archet, Nice
  - CHR d'Orléans Hopital la Source, Orléans
  - Hopital St Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hopital Tenon, Paris
  - CH Francois Miterrand, Pau
  - CH Poissy, Poissy
  - CH de Pontoise, Pontoise
  - CH de la Région d'Annecy, Pringy
  - CH Leon Binet, Provins
  - CH de St-Brieuc, Saint-Brieuc
  - Hopital Delafontaine, Saint-Denis
  - HIA Béjin, Saint-Mandé
  - CH de St-Malo, St-Malo
  - CHRU Bretonneau, Tours
  - Hopital Jean Bernard, Valenciennes
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Payen JF, Chanques G, Mantz J, Hercule C, Auriant I, Leguillou JL, Binhas M, Genty C, Rolland C, Bosson JL. Current practices in sedation and analgesia for mechanically ventilated critically ill patients: a prospective multicenter patient-based study. Anesthesiology. 2007 Apr;106(4):687-95; quiz 891-2. doi: 10.1097/01.anes.0000264747.09017.da. PMID 17413906
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Constantin JM, Chanques G, De Jonghe B, Sanchez P, Mantz J, Payen JF, Sztark F, Richebe P, Lagneau F, Capdevila X, Bazin JE, Lefrant JY. [Current use of sedation and analgesia: 218 resuscitations in France services practices survey]. Ann Fr Anesth Reanim. 2010 May;29(5):339-46. doi: 10.1016/j.annfar.2010.01.014. Epub 2010 Apr 13. French. PMID 20392591
- [Background] Brook AD, Ahrens TS, Schaiff R, Prentice D, Sherman G, Shannon W, Kollef MH. Effect of a nursing-implemented sedation protocol on the duration of mechanical ventilation. Crit Care Med. 1999 Dec;27(12):2609-15. doi: 10.1097/00003246-199912000-00001. PMID 10628598
- [Background] De Jonghe B, Bastuji-Garin S, Fangio P, Lacherade JC, Jabot J, Appere-De-Vecchi C, Rocha N, Outin H. Sedation algorithm in critically ill patients without acute brain injury. Crit Care Med. 2005 Jan;33(1):120-7. doi: 10.1097/01.ccm.0000150268.04228.68. PMID 15644658
- [Background] Quenot JP, Ladoire S, Devoucoux F, Doise JM, Cailliod R, Cunin N, Aube H, Blettery B, Charles PE. Effect of a nurse-implemented sedation protocol on the incidence of ventilator-associated pneumonia. Crit Care Med. 2007 Sep;35(9):2031-6. doi: 10.1097/01.ccm.0000282733.83089.4d. PMID 17855817
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- [Background] Treggiari MM, Romand JA, Yanez ND, Deem SA, Goldberg J, Hudson L, Heidegger CP, Weiss NS. Randomized trial of light versus deep sedation on mental health after critical illness. Crit Care Med. 2009 Sep;37(9):2527-34. doi: 10.1097/CCM.0b013e3181a5689f. PMID 19602975
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Derived] SRLF Trial Group. Impact of oversedation prevention in ventilated critically ill patients: a randomized trial-the AWARE study. Ann Intensive Care. 2018 Sep 21;8(1):93. doi: 10.1186/s13613-018-0425-3. PMID 30242747